CLINICAL TRIAL: NCT04314271
Title: The Observational Study of Cardiac and Pulmonary Ultrasound and Evaluation of Treatment of Severe Patients With Novel Coronavirus Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202003028
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Novel Coronavirus Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Complete the examination of cardio-pulmonary ultrasound in accordance with the a-ccue process of patients with novel coronavirus bedside. To summarize and analyze the characteristics of cardiopulmonary ultrasound in patients with novel coronavirus pneumonia, and assess the relationship between pulmonary ultrasound imaging score and National Early Warning Score(NEWS) and prognosis. Auto line B is a method which is based on artificial intelligence is used to calculate the lungs ultrasonic B line numbers reviewing the status of patients with lung, and also evaluate patients' lungs using the traditional artificial semi-quantitative method, to evaluate those two kinds of evaluation methods for the evaluation of patients with lung condition effects are consistent or not, and verify consistency of ultrasonic evaluation method and the way of CT evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. age >18 years old
2. identify the patients infected with novel coronavirus pneumonia;
3. the patient completed CT examination;
4. sign the informed consent.

Exclusion Criteria:

1. age < 18;
2. those who cannot complete cardiopulmonary ultrasound according to the a-ccue process;
3. the patient or his guardian requests to withdraw from the researcher;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (Age ≥ 18 years) patients with novel coronavirus pneumonia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-20 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
characteristics of cardiopulmonary ultrasound | 30 mins
  Complete the examination of cardio-pulmonary ultrasound in accordance with the a-ccue process of patients with novel coronavirus bedside. To summarize and analyze the characteristics of cardiopulmonary ultrasound in patients with novel coronavirus pneumonia

SECONDARY OUTCOMES:
assess the relationship between pulmonary ultrasound imaging score and National Early Warning Score(NEWS) and prognosis. | 2-3weeks
  assess the relationship between pulmonary ultrasound imaging score and National Early Warning Score(NEWS) and prognosis.

OTHER OUTCOMES:
evaluate two kinds of evaluation methods for the evaluation of patients with lung condition effects are consistent or not, and verify consistency of ultrasonic evaluation method and the way of CT evaluation. | 3 hours
  Auto line B is a method which is based on artificial intelligence is used to calculate the lungs ultrasonic B line numbers reviewing the status of patients with lung, and also evaluate patients' lungs using the traditional artificial semi-quantitative method, to evaluate those two kinds of evaluation methods for the evaluation of patients with lung condition effects are consistent or not

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Li Na, MD, Study Chair — Xiangya Hospital
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China